CLINICAL TRIAL: NCT05939167
Title: A Double-blind, Randomized Placebo-controlled Clinical Trial to Investigate the Safety and Efficacy of Mesenchymal Stem Cells Treatment for AIDS Patients at Late Stage
Brief Title: Mesenchymal Stem Cells Treatment for AIDS Patients at Late Stage
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cell Energy Life Sciences Group Co. LTD (Industry)
Collaborators: Beijing 302 Hospital (Other); Shenzhen Third People's Hospital (Other); Fifth Hospital of Shijiazhuang City (Other); Beijing YouAn Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022YFC2304403
Record Dates: First submitted 2023-05-15; First posted 2023-07-11 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- placebo control (Placebo Comparator): use saline
  Interventions: Other: saline
- mesenchymal stem cells standard treatment (Experimental): transplant mesenchymal stem cells for 3 times
  Interventions: Drug: mesenchymal stem cell
- mesenchymal stem cells enhanced treatment (Experimental): transplant mesenchymal stem cells for 6 times

INTERVENTIONS:
Drug: mesenchymal stem cell — Mesenchymal stem cell dose is 0.75-1.0×10*6/kg and is transplanted by intravenous infusion. For the mesenchymal stem cell standard treatment group, the cells are used for three times(at week 0, 2,4 after recruitment) and the mesenchymal stem cell enhanced treatment group, the cells are used for six times(at week 0, 2,4,24,26,28 after recruitment).
  Other Names: umbilical cord derived MSCs
  Arms: mesenchymal stem cells standard treatment
Other: saline — saline is used as placebo in the placebo comparator group
  Arms: placebo control

SUMMARY:
The goal of this study is to conduct a prospective, double-blind, randomized placebo-controlled clinical trial to investigate the safety and efficacy of mesenchymal stem cells treatment for AIDS patients at late stage.

DETAILED DESCRIPTION:
Mesenchymal stem cells (MSCs) possess immunomodulatory, anti-inflammatory, and regenerative properties. The safety and effectiveness of MSCs have been investigated in various clinical trials for the treatment of several disorders, including graft-versushost disease, inflammatory bowel disease, and multiple sclerosis. It has been reported that MSC treatment in HIV-infected patients with immunological nonresponders resulted in a significant increase in circulating CD4+ T lymphocytes and a decrease of the activation of T lymphocytes and soluble inflammation mediator levels without significant adverse effects or loss of viremia control. However, the therapeutic efficacy of MSC treatment for AIDS patients at late stage is not well-understood. This study aims to investigate the safety and efficacy of MSC treatment for AIDS patients at late stage.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV infection, aged 18-65, both genders
2. CD4+T count less than 500 cells/ul at baseline.
3. No serious AIDS related events. 3. could understand and sign the informed consent form and comply with the requirements of this study.

4. agree not to participate in other studies and not to receive other immunotherapies during the period of participation in this study

Exclusion Criteria:

1. have HBV/HCV/HDV/HEV infection, and the virological test is positive.
2. The viral load for CMV and EBV is more than 1000 copies/ML.
3. have HIV-2 infection.
4. have serious complications in organs including renal, circulatory, respiratory, digestive, endocrine, neural and immunological diseases and tumors.
5. received treatment of hormones or other immunosuppressive drugs for a long time.
6. with serious AIDS related or unrelated events.
7. received immunosuppressive drugs or systemic cytotoxic drugs for more than 3 months before recruiting
8. have poor compliance during treatment.
9. drug addiction within 6 months, or the urine drug test is positive
10. participate in other clinical trials currently
11. pregnant, breastfeeding, or have fertility requirements.
12. unable or unwilling to provide informed consents, or unable to comply with research requirements.
13. Other serious situations that may hinder clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2027-07-10 (Estimated); Study Completion 2028-07-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with side effects in MSCs treatment groups | 48 weeks
  Investiagte the number of participants with treatment-related adverse events as assessed by CTCAE v4.0 after MSCs infusion.
CD4+ T cell counts after MSCs transfusion | 48 weeks
  at week 12, 24 and 48, evaluate CD4+ T cell counts and compare with baseline

SECONDARY OUTCOMES:
HIV RNA viral load | 48 weeks
  At week 12, 24 and 48, test HIV RNA viral load in participants' blood using RT-PCR and compare with baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, Doctor, Principal Investigator — Beijing 302 Hospital
Locations (4):
- China (4):
  - Beijing 302 Hospital, Beijing
  - Beijing YouAn Hospital, Beijing
  - Shenzhen Third People's Hospital, Shenzhen
  - The Fifth Hospital of Shijiazhuang, Shijiazhuang

IPD SHARING:
Plan to Share IPD: No